CLINICAL TRIAL: NCT00102479
Title: A Phase II Study to Test PK Tolerability in Children and Adolescents
Brief Title: Aripiprazole Pharmacokinetics (PK) and Tolerability Study in Children and Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: 31-03-238
Record Dates: First submitted 2005-01-29; First posted 2005-01-31 (Estimated); Last update posted 2006-04-17 (Estimated); Status verified 2006-04

CONDITIONS: Schizophrenia; Mania
Keywords: Pharmacokinetics,; Aripiprazole; acute mania in pediatric populations
MeSH Terms: conditions — Schizophrenia; Mania | interventions — Aripiprazole

INTERVENTIONS:
Drug: Aripiprazole

SUMMARY:
The purpose of this trial is to assess the safety, tolerability and pharmacokinetics of aripiprazole tablets following oral administration to children and adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents between 10-17 years, in good physical health, preferentially with a primary schizophrenia spectrum diagnosis or bipolar spectrum disorder

Exclusion Criteria:

* History of mental retardation
* Any neurological disorder with the exception of Pervasive Developmental Disorder (PDD), Attention Deficit Hyperactivity Disorder (ADHD), and Tourette's Syndrome

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2004-07; Study Completion 2005-07

REFERENCES:
- [Derived] Findling RL, Kauffman RE, Sallee FR, Carson WH, Nyilas M, Mallikaarjun S, Shoaf SE, Forbes RA, Boulton DW, Pikalov A. Tolerability and pharmacokinetics of aripiprazole in children and adolescents with psychiatric disorders: an open-label, dose-escalation study. J Clin Psychopharmacol. 2008 Aug;28(4):441-6. doi: 10.1097/JCP.0b013e31817dd520. PMID 18626272